CLINICAL TRIAL: NCT06850103
Title: A Phase II Exploratory Multicenter Randomized Controlled Clinical Trial to Evaluate the Effectiveness of Neoadjuvant Short-Course Radiotherapy (SCRT) Followed by CAPEOX Chemotherapy and Serplulimab in Microsatellite Stable (MSS) or Proficient Mismatch Repair (pMMR) Rectal Cancer With Synchronous Oligometastases
Brief Title: SCRT-CAPEOX-Serplulimab for MSS/pMMR Rectal Cancer With Oligometastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Ningbo No.2 Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Second Affiliated Hospital of Wenzhou Medical University (Other); Ningbo No. 1 Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); The Affiliated People's Hospital of Ningbo University (Other Government)
Responsible Party: Principal Investigator, Feng Ye, chief physician, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRT-CAP-Serp TriFire
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Carcinoma; Oligometastases; pMMR; MSS; iTNT
MeSH Terms: conditions — Colorectal Neoplasms | interventions — XELOX; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients in the experimental arm will receive short-course radiotherapy (SCRT) followed by 4 cycles of CAPEOX chemotherapy plus Serplulimab as neoadjuvant therapy, then undergo TME resection of the primary tumor and local treatment of metastatic lesions, followed by 4 additional cycles of CAPEOX plus Serplulimab as adjuvant therapy.
  Interventions: Radiation: short-course radiotherapy; Drug: CAPEOX/XELOX; Drug: Serplulimab; Procedure: surgery
- Active Comparator (Active Comparator): Patients in the control arm will receive short-course radiotherapy (SCRT) followed by 4 cycles of CAPEOX chemotherapy as neoadjuvant therapy, then undergo TME resection of the primary tumor and local treatment of metastatic lesions, followed by 4 additional cycles of CAPEOX as adjuvant therapy.
  Interventions: Radiation: short-course radiotherapy; Drug: CAPEOX/XELOX; Procedure: surgery

INTERVENTIONS:
Radiation: short-course radiotherapy — Neoadjuvant short-course radiotherapy (SCRT) will be administered at a total dose of 25 Gy, delivered in 5 fractions of 5 Gy each.
Drug: CAPEOX/XELOX — Capecitabine: 1000 mg/m² BID, D1-14, Q3W × 4 cycles Oxaliplatin: 130 mg/m² IV, D1, Q3W × 4 cycles
Drug: Serplulimab — Serplulimab: 300 mg IV, D1, Q3W × 4 cycles
  Arms: Experimental
Procedure: surgery — Primary tumor: Total Mesorectal Excision (TME) Metastatic lesions: Local therapeutic intervention

SUMMARY:
Background and Significance:

Colorectal cancer (CRC) ranks as the third most common cancer and the second leading cause of cancer-related deaths globally. Despite improved early screening rates, a significant proportion of newly diagnosed CRC patients present with synchronous metastases, predominantly liver metastases. The concept of oligometastases, introduced by Hellman and Weichselbaum in 1995, describes a transitional state between localized disease and widespread metastases, characterized by limited metastatic lesions (typically 1-5) confined to 1-2 organs.

Current Treatment Landscape:

The management of oligometastatic disease combines local therapeutic approaches (surgery, radiotherapy, radiofrequency ablation) with systemic treatments, aiming to achieve No Evidence of Disease (NED) status. The ESMO guidelines officially categorized metastatic CRC into oligometastatic and widespread metastatic states in 2016, emphasizing the importance of integrated local and systemic treatments for oligometastatic colorectal liver metastases (CRLM).

Treatment Evolution and Challenges:

While the EPOC study established CAPEOX neoadjuvant chemotherapy followed by R0 resection as the standard treatment for initially resectable CRLM, patients with synchronous rectal cancer oligometastases present unique challenges due to complex local anatomy and high local recurrence risks. Although various neoadjuvant approaches, including Total Neoadjuvant Therapy (TNT), have been studied, they have not demonstrated significant long-term survival benefits, primarily because distant metastases impact survival more significantly than local recurrence.

Innovative Approach:

Recent success with Immunotherapy-Based Total Neoadjuvant Therapy (iTNT) in microsatellite stable/proficient mismatch repair (MSS/pMMR) locally advanced rectal cancer has shown promising results. Short-course radiotherapy (SCRT) combined with chemotherapy and immunotherapy has demonstrated superior efficacy trends, attributed to radiation's immune-activating effects on both local and distant tumor microenvironments.

Research Objective:

This project aims to evaluate the effectiveness of iTNT combined with SCRT in MSS/pMMR rectal cancer patients with synchronous oligometastases. The novel approach integrates SCRT with CAPEOX chemotherapy and Serplulimab, potentially improving complete response rates, organ preservation opportunities, and overall treatment efficacy while reducing recurrence risks. This pioneering study represents the first investigation of iTNT in synchronous rectal cancer oligometastases, offering a potentially transformative treatment strategy for this challenging patient population.

Research Innovation:

The study uniquely combines SCRT, CAPEOX chemotherapy, and Serplulimab in a neoadjuvant setting for MSS/pMMR synchronous rectal cancer oligometastases, addressing an unmet clinical need and potentially establishing a new treatment paradigm in this field.

ELIGIBILITY:
Inclusion Criteria:

- Has signed the written Informed Consent Form (ICF) and is able to comply with protocol-specified visits and procedures.

Age between 18-75 years.

Histologically confirmed primary rectal adenocarcinoma, with MRI showing tumor location within 10cm from the anal verge.

Synchronous oligometastatic rectal cancer confirmed by comprehensive imaging evaluation (contrast-enhanced CT, contrast-enhanced MRI, PET-CT, etc.), with ≤2 metastatic sites and ≤5 total metastatic lesions.

Microsatellite stability status confirmed as MSS (using the NCI-recommended 5 microsatellite markers: BAT25, BAT26, D5S346, D2S123, D17S250) or proficient mismatch repair (pMMR) status confirmed by immunohistochemistry showing positive nuclear expression of all 4 MMR proteins (MLH1, MSH2, MSH6, PMS2).

At least one measurable lesion according to RECIST v1.1 criteria.

Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1.

Adequate organ function and bone marrow reserve, defined as follows:

Complete blood count:

Absolute Neutrophil Count (ANC) ≥1.5×109/L Platelet count (PLT) ≥100×109/L Hemoglobin (HGB) ≥10.0g/dL

Liver function:

Total Bilirubin (TBIL) ≤1.5×Upper Limit of Normal (ULN) Alanine transaminase (ALT) and Aspartate aminotransferase (AST) ≤3×ULN Serum albumin (ALB) ≥35 g/L

Renal function:

Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min (calculated using Cockcroft-Gault formula [see Appendix 3] or standard 24-hour urine collection method) Urine protein by dipstick <2+ For subjects with baseline urine protein ≥2+ by dipstick, 24-hour urine protein must be <1g

Coagulation:

International Normalized Ratio (INR) ≤1.5 Activated partial thromboplastin time (APTT) ≤1.5×ULN Certain anticoagulant medications (such as antiplatelet agents, vitamin K antagonists) must be discontinued 7-14 days before surgery and replaced with alternative medications (such as low molecular weight heparin) No concurrent serious diseases that would threaten subject survival (leading to expected survival <5 years).

Women of childbearing potential and men whose partners are of childbearing potential must use effective contraception during the entire treatment period and for 6 months after treatment completion. Female subjects must either have evidence of post-menopausal status, or if pre-menopausal, have a negative urine or serum pregnancy test.

Exclusion Criteria:

- More than 2 metastatic sites or more than 5 total metastatic lesions confirmed by imaging evaluation.

Prior anti-tumor therapy for the study disease, including surgery, radiotherapy, chemotherapy, targeted therapy, or immunotherapy.

Previous treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies, or any other drugs targeting T-cell co-stimulation or immune checkpoint pathways (e.g., OX40, CD137), or adoptive cell immunotherapy.

Concurrent participation in another clinical trial, except for observational (non-interventional) studies or survival follow-up phase of interventional studies.

Receipt of any investigational drug within 4 weeks prior to first dose of study drug.

History of blood transfusion or use of G-CSF, GM-CSF, EPO, TPO, or IL-11 within 14 days prior to screening laboratory tests.

Use of immunosuppressive medications within 4 weeks prior to first dose of study drug, excluding:

Intranasal inhaled corticosteroids or local steroid injections Systemic corticosteroids at ≤10 mg/day prednisone equivalent Corticosteroids as premedication for allergic reactions (e.g., CT contrast) Traditional Chinese medicines with anti-tumor indications or immunomodulatory effects within 1 week prior to first dose Receipt of live or attenuated vaccines within 4 weeks prior to first dose or anticipated during the study period.

Major surgery within 4 weeks prior to first dose (e.g., craniotomy, thoracotomy, or laparotomy), anticipated major surgery during treatment (excluding protocol-specified rectal cancer surgery), or presence of unhealed wounds, ulcers, or fractures.

Known active or suspected autoimmune disease or history within past 2 years (exceptions: eczema, vitiligo, psoriasis, alopecia, or Graves' disease not requiring systemic treatment in past 2 years; hypothyroidism requiring only hormone replacement; Type I diabetes requiring only insulin).

Known history of primary immunodeficiency.

Active tuberculosis, current anti-TB treatment, or anti-TB treatment within 1 year prior to first dose.

Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

Known allergy to capecitabine, oxaliplatin, serplulimab, or other monoclonal antibody components.

Clinically significant ascites, pleural effusion requiring intervention, or symptomatic pericardial effusion requiring drainage.

HIV infection (HIV antibody positive).

Acute or chronic active hepatitis B (defined as HBsAg positive or HBcAb positive only with HBV DNA ≥2000 IU/mL or ≥1×104 copies/mL) or hepatitis C (defined as HCV antibody positive with detectable HCV RNA).

Active syphilis infection requiring treatment.

Severe infection within 4 weeks prior to first dose, including but not limited to hospitalization for infection, bacteremia, or severe pneumonia; therapeutic oral or IV antibiotics within two weeks prior to first dose.

Symptomatic congestive heart failure (NYHA class II-IV) or LVEF <50%; symptomatic or uncontrolled arrhythmias; congenital long QT syndrome or QTc >500 ms at screening (Fridericia's formula).

Uncontrolled hypertension (SBP ≥160 mmHg or DBP ≥100 mmHg) despite standard therapy, history of hypertensive crisis or encephalopathy.

Severe bleeding diathesis or coagulation disorders, or current thrombolytic therapy.

Any arterial thromboembolic events within 6 months prior to first dose, including myocardial infarction, unstable angina, stroke, or TIA.

Esophageal or gastric varices requiring immediate intervention; high bleeding risk subjects require endoscopic evaluation within 3 months before enrollment.

History of GI perforation and/or fistula within 6 months prior to first dose.

Life-threatening bleeding event within 3 months prior to first dose, or Grade 3/4 GI/variceal bleeding requiring transfusion, endoscopy, or surgery.

History of DVT, PE, or other serious thromboembolism within 3 months prior to first dose (excluding catheter-related thrombosis or superficial thrombosis).

Uncontrolled metabolic disorders or other non-malignant conditions causing high medical risk or uncertain survival evaluation.

Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh B >7 or worse cirrhosis.

Bowel obstruction (including incomplete requiring parenteral nutrition); conditions with perforation risk; history of extensive bowel resection, Crohn's disease, ulcerative colitis, or chronic diarrhea.

Interstitial lung disease requiring treatment; history of pulmonary fibrosis, pneumoconiosis, drug-induced pneumonitis, organizing pneumonia, or severe pulmonary dysfunction.

Significant malnutrition (5% weight loss within 1 month or 15% within 3 months of consent, or >50% reduced intake for 1 week), unless corrected for ≥4 weeks before first dose.

History of other primary malignancies, except:

Cured malignancies with ≥2 years disease-free and low recurrence risk Well-treated non-melanoma skin cancer or lentigo maligna Well-treated carcinoma in situ

Other acute or chronic conditions that could:

Increase study participation risks Interfere with result interpretation Make subject unsuitable per investigator judgment Neurological, psychiatric, or social conditions affecting compliance or safety assessment.

Alcohol, drug, or substance abuse affecting drug administration or toxicity analysis.

Pregnant or breastfeeding women.

Conditions interfering with medication management or toxicity analysis due to alcohol, drug, or substance use.

Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
3-year PFS | within 3 years from study enrollment.

SECONDARY OUTCOMES:
No Evidence of Disease (NED) rate | Within 3 months after surgery
Primary tumor pathological complete response (pCR) rate | After surgery
3-year local recurrence rate (LRR) | within 3 years after primary treatment
5-year OS | within 5 years from study enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No